CLINICAL TRIAL: NCT00494091
Title: Phase 2, Non Randomized, Open Label Study Of Temsirolimus (CCI-779) In Subjects With Advanced Renal Cell Carcinoma (RCC)
Brief Title: Study Evaluating The Safety, Efficacy & Pharmacokinetics Of Temsirolimus(CCI-779) In Subjects With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-2217; B1771002
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. (Experimental)
  Interventions: Drug: Temsirolimus (CCI-779)
- B. (Experimental)
  Interventions: Drug: Temsirolimus (CCI-779)

INTERVENTIONS:
Drug: Temsirolimus (CCI-779) — 20 mg/m2 IV TEMSR weekly (Japan, n=6)
  Other Names: Torisel
  Arms: A.
Drug: Temsirolimus (CCI-779) — 25 mg IV TEMSR weekly (all other pts)
  Other Names: Torisel
  Arms: B.

SUMMARY:
This is a study to evaluate the safety, efficacy and pharmacokinetics of temsirolimus in Asian patients with advanced renal cell carcinoma. The trial is only being conducted in Japan, Korea, and China.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed, advanced (stage IV or recurrent disease) RCC. The American Joint Committee on Cancer (AJCC) staging and classification criteria will be used.
* ECOG performance status of 0-1.
* At least one measurable lesion per RECIST.
* Age greater than or equal to 20 years.
* Japanese, Chinese, or Korean ethnicity.

Exclusion Criteria:

* CNS metastases at screening or history or CNS metastases.
* Prior targeted, chemotherapeutic, cytokine-based, or other investigational agents for the treatment of RCC within 4 weeks before first dose of test article. Subjects must have documented objective progressive disease after any prior systemic RCC treatment and have recovered to grade 1 or lower toxicities from effects of prior systemic therapy for RCC.
* In past 5 years, other prior malignancy (except basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- China (3):
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- Japan (14):
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Gunma
  - Pfizer Investigational Site, Hokkaido
  - Pfizer Investigational Site, Ibaraki
  - Pfizer Investigational Site, Kagawa
  - Pfizer Investigational Site, Kagoshima
  - Pfizer Investigational Site, Kyoto
  - Pfizer Investigational Site, Nara
  - Pfizer Investigational Site, Okayama
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Shizuoka
  - Pfizer Investigational Site, Tokyo
  - Pfizer Investigational Site, Yamagata
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-2217&StudyName=Study%20Evaluating%20The%20Safety%2C%20Efficacy%20%26%20Pharmacokinetics%20Of%20Temsirolimus%28CCI-779%29%20In%20Subjects%20With%20Advanced%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Temsirolimus 20 mg/m^2: Temsirolimus 20 milligrams per square meter (mg/m^2) intravenously (IV) once weekly until disease progression, unacceptable toxicity, or withdrawal of consent.
- Temsirolimus 25 mg: Temsirolimus 25 mg IV once weekly until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Overall Study
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Started | 6 | 76
Completed | 0 | 0
Not Completed | 6 | 76
Not completed — Death | 5 | 54
Not completed — Lost to Follow-up | 0 | 4
Not completed — Other | 1 | 11
Not completed — Withdrawal by Subject | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg | Total
Number analyzed (Participants) | 6 | 76 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 59.67 (10.29) | 55.20 (11.52) | 55.52 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 23 | 23
  Male | 6 | 53 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit: confirmed complete response (CR) or partial response (PR) or had stable disease (SD) lasting at least 24 weeks. CR was the disappearance of all target lesions and nontarget lesions. PR was at least a 30 percent (%) decrease in sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. SD was having neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Time Frame: Baseline Up to 4 years
Population: Intent-to-treat (ITT) population included all participants who were enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Number analyzed (Participants) | 6 | 76
percentage of participants | 50.0 [11.8 to 88.2] | 48.7 [37.0 to 60.4]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Median time from the date of enrollment to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: Baseline Up to 4 years
Population: ITT population included all participants who were enrolled in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Number analyzed (Participants) | 6 | 76
months | 8.7 [4.0 to 29.0] | 7.3 [3.8 to 9.9]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR according to Response Evaluation Criteria In Solid Tumors (RECIST). CR is disappearance of all target lesions. PR shows at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Baseline Up to 4 years
Population: ITT population included all participants who were enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Number analyzed (Participants) | 6 | 76
percentage of participants | 0 [0 to 0] | 11.8 [5.6 to 21.3]

4. Secondary Outcome: Duration of Response
Description: Time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest sum longest diameters (LD) recorded since enrollment.
Time Frame: Baseline Up to 4 years
Population: Intent-to-treat ITT population included all participants who were enrolled in this study. Here N (number of participants analyzed) signifies participants with objective disease response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Number analyzed (Participants) | 0 | 9
months |  | 31.3 [4.5 to NA] — The upper limit of 95 percent (%)confidence interval (CI) is not available because there was no recurrence observation after median.

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from the date of enrollment to the date of the first documentation of PD, the date of treatment discontinuation except completion of treatment, or date of death due to cancer.
Time Frame: Baseline Up to 4 years
Population: ITT population included all participants who were enrolled in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Number analyzed (Participants) | 6 | 76
months | 7.7 [1.9 to 29.0] | 5.4 [3.5 to 7.4]

6. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the date of enrollment to date of death due to any cause. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline Until Death (Up to 4 years)
Population: ITT population included all participants who were enrolled in this study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Temsirolimus 25 mg IV: Temsirolimus 25 mg IV once weekly until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg IV
Number analyzed (Participants) | 6 | 76
months | 29.1 [4.4 to 36.3] | 17.8 [13.5 to 25.3]

7. Other Pre Specified Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Sirolimus is a major metabolite of temsirolimus. As per planned analysis, only participants in "Temsirolimus 20 mg/m^2" treatment arm were to be drawn blood samples intensively for pharmacokinetic analysis.
Time Frame: 0 hours (pre-dose), 0.5 hours, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study treatment and had at least 3 measurable blood concentration samples available. Here N (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL)
  Cmax for temsirolimus at Week 1 | 704 (207)
  Cmax for temsirolimus at Week 4 | 640 (308)
  Cmax for sirolimus at Week 1 | 69.6 (13.1)
  Cmax for sirolimus at Week 4 | 83.0 (38.0)

8. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: as for outcome 7
Time Frame: 0 hours (pre-dose), 0.5, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: PK population included all participants who received at least 1 dose of study treatment and had at least 3 measurable blood concentration samples available. Here N (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
hours
  Tmax for temsirolimus | 0.50 [0.50 to 0.58]
  Tmax for sirolimus | 2.0 [2.0 to 24.0]

9. Other Pre Specified Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Sirolimus is the major metabolite of temsirolimus. As per planned analysis, only participants in "Temsirolimus 20 mg/m^2" treatment arm were to be drawn blood samples intensively for pharmacokinetic analysis.
Time Frame: 0 hours (pre-dose), 0.5, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
hours
  t1/2 for temsirolimus at Week 1 | 18.6 (6.5)
  t1/2 for temsirolimus at Week 4 | 18.2 (5.43)
  t1/2 for sirolimus at Week 1 | 54.7 (15.2)
  t1/2 for sirolimus at Week 4 | 52.4 (12.4)

10. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUC)
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Sirolimus is the major metabolite of temsirolimus. As per planned analysis, only participants in "Temsirolimus 20 mg/m^2" treatment arm were to be drawn blood samples intensively for pharmacokinetic analysis.
Time Frame: 0 hours (pre-dose), 0.5 hours, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
ng*h/mL
  AUC for temsirolimus at Week 1 | 2819 (1065)
  AUC for temsirolimus at Week 4 | 2163 (822)
  AUC for sirolimus at Week 1 | 6902 (3127)
  AUC for sirolimus at Week 4 | 5582 (3420)

11. Other Pre Specified Outcome: Clearance (CLss) of Temsirolimus
Description: Steady state total body clearance equals infusion rate (zero order) divided by steady state plasma concentration of temsirolimus (R0/Css). As per planned analysis, only participants in "Temsirolimus 20 mg/m^2" treatment arm were to be drawn blood samples intensively for pharmacokinetic analysis.
Time Frame: 0 hours (pre-dose), 0.5, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
Liter per hour (L/h)
  Week 1 | 13.6 (4.74)
  Week 4 | 17.1 (5.71)

12. Other Pre Specified Outcome: Volume of Distribution at Steady State (Vss) of Temsirolimus
Description: Vss is an estimate of the volume of distribution at steady state. It is used to predict the plasma concentrations following multiple dosing to a steady-state or pseudo-equilibrium. Vss is proportional to the amount of drug in the body versus the plasma concentration of the drug at steady state. As per planned analysis, only participants in "Temsirolimus 20 mg/m^2" treatment arm were to be drawn blood samples intensively for pharmacokinetic analysis.
Time Frame: 0 hours (pre-dose), 0.5, 1, 2, 6, 24, 72, and 96 hours during Week 1 and 4 of treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Temsirolimus 20 mg/m^2
Number analyzed (Participants) | 5
Liter
  Week 1 | 243 (64.7)
  Week 4 | 250 (75.7)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Temsirolimus 20 mg/m^2 | Temsirolimus 25 mg
Serious Adverse Events (participants affected / at risk) | 4/6 | 28/76
Other Adverse Events (participants affected / at risk) | 6/6 | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 20 mg/m^2 (N=6) | Temsirolimus 25 mg (N=76)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 6
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Circulatory collapse (Vascular disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 20 mg/m^2 (N=6) | Temsirolimus 25 mg (N=76)
Anaemia (Blood and lymphatic system disorders) | 5 | 23
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 7
Lymphopenia (Blood and lymphatic system disorders) | 2 | 8
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 9
Palpitations (Cardiac disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 9
Abdominal distension (Gastrointestinal disorders) | 0 | 6
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 4
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 3 | 17
Dental caries (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 17
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 3
Glossitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 9
Nausea (Gastrointestinal disorders) | 0 | 18
Periodontitis (Gastrointestinal disorders) | 1 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 1
Radicular cyst (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 42
Toothache (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 11
Asthenia (General disorders) | 0 | 10
Axillary pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 6
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 1 | 6
Face oedema (General disorders) | 1 | 9
Fatigue (General disorders) | 3 | 25
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 2
Generalised oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 5
Localised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 13
Pyrexia (General disorders) | 3 | 28
Thirst (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 3
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Nail infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 8
Onychomycosis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 0 | 7
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Rash pustular (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 2
Sputum purulent (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 20
Urinary tract infection (Infections and infestations) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 5 | 23
Aspartate aminotransferase increased (Investigations) | 5 | 23
Bacterial test positive (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 3 | 3
Blood alkaline phosphatase (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 4 | 12
Blood calcium decreased (Investigations) | 2 | 3
Blood magnesium increased (Investigations) | 1 | 0
Blood chloride increased (Investigations) | 0 | 2
Blood cholesterol increased (Investigations) | 2 | 12
Blood creatine increased (Investigations) | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood creatinine (Investigations) | 0 | 4
Blood creatinine increased (Investigations) | 2 | 20
Blood glucose increased (Investigations) | 0 | 9
Blood iron decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase (Investigations) | 0 | 2
Blood lactate dehydrogenase decreased (Investigations) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 3 | 13
Blood phosphorus decreased (Investigations) | 1 | 2
Blood potassium decreased (Investigations) | 1 | 2
Blood potassium increased (Investigations) | 1 | 2
Blood pressure increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 2
Blood triglycerides increased (Investigations) | 3 | 16
Blood urea (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 4
C-reactive protein increased (Investigations) | 2 | 2
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 7
Glycosylated haemoglobin increased (Investigations) | 2 | 7
Haematocrit decreased (Investigations) | 0 | 5
Haemoglobin (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 23
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 6
Neutrophil count increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 3 | 18
Platelet count increased (Investigations) | 1 | 3
Protein total decreased (Investigations) | 1 | 1
Protein total increased (Investigations) | 1 | 4
Prothrombin time prolonged (Investigations) | 4 | 0
Pulmonary function test abnormal (Investigations) | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 4
Red blood cell count increased (Investigations) | 0 | 2
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 5 | 18
Weight increased (Investigations) | 0 | 4
White blood cell count decreased (Investigations) | 0 | 14
White blood cell count increased (Investigations) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 35
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 34
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 28
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 4
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 7
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 31
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 8
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 28
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 5
Dysgeusia (Nervous system disorders) | 3 | 7
Headache (Nervous system disorders) | 1 | 6
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Parosmia (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Breath holding (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 8
Azotaemia (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 3
Polyuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 4
Testicular swelling (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 15
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 12
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 20
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 7
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 23
Rash (Skin and subcutaneous tissue disorders) | 6 | 43
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 11
Phlebitis (Vascular disorders) | 1 | 2
Cardiac valve disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 3
Breath odour (Gastrointestinal disorders) | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Chest X-ray abnormal (Investigations) | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 3
Spinal cord compression (Nervous system disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.